CLINICAL TRIAL: NCT01965535
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination for 12 Weeks With Ribavirin or for 24 Weeks Without Ribavirin in Treatment-Experienced Cirrhotic Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination ± Ribavirin in Cirrhotic Subjects With Chronic Genotype 1 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-337-0121; 2013-002296-17 (EudraCT Number)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-06

CONDITIONS: HCV Infection
Keywords: Hepatitis C; HCV; Cirrhosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDV/SOF (Experimental): LDV/SOF FDC tablet plus placebo to match RBV for 24 weeks
  Interventions: Drug: LDV/SOF; Drug: Placebo to match RBV
- LDV/SOF + RBV (Experimental): Placebo to match SOF/LDV FDC plus placebo to match RBV for 12 weeks, followed by LDV/SOF FDC plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV; Drug: Placebo to match LDV/SOF; Drug: Placebo to match RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF (90/400 mg) FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
Drug: RBV — RBV (200 mg tablets) administered orally in a divided daily dose based on weight (1000 mg per day for participants weighing < 75 kg; 1200 mg per day for participants weighing ≥ 75 kg)
  Arms: LDV/SOF + RBV
Drug: Placebo to match LDV/SOF — Placebo to match LDV/SOF administered orally once daily
  Arms: LDV/SOF + RBV
Drug: Placebo to match RBV — Placebo to match RBV administered orally in a divided daily dose

SUMMARY:
This study is to determine the antiviral efficacy of sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) with and without ribavirin (RBV), and to evaluate the safety and tolerability of each regimen as assessed by review of the accumulated safety data. Approximately 150 participants with genotype 1 HCV infection, who have previously received treatment for HCV, and who have a diagnosis for cirrhosis will be enrolled. Participants will be randomized to 1 of 2 groups.

Group 1: SOF/LDV FDC tablet plus placebo to match RBV for 24 weeks

Group 2: Delayed treatment group: placebo to match SOF/LDV FDC plus placebo to match RBV for 12 weeks, followed by SOF/LDV FDC once daily plus RBV in a divided daily dose for 12 weeks

Randomization will 1:1 to the two groups and will be stratified by HCV genotype (1a, 1b; mixed or other genotype 1 results will be stratified as genotype 1a), and prior HCV therapy treatment response (never achieved HCV RNA < the lower limit of quantitation (LLOQ), or achieved HCV RNA < LLOQ).

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years, with chronic genotype 1 HCV infection
* HCV RNA ≥ 10,000 IU/mL at screening
* Prior virological failure after treatment with pegylated interferon (PEG-IFN), RBV and a protease inhibitor following documented prior virology failure after treatment with a PEG-IFN + RBV regimen
* Evidence of cirrhosis
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* Prior exposure to approved or experimental HCV specific direct-acting antivirals other than a nonstructural protein (NS)3/4A protease inhibitor
* History of solid organ transplantation, including liver transplant
* Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Hyland, DPhil, Study Director — Gilead Sciences
Locations (16):
- France (16):
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Montpelier
  - Nancy
  - Nice
  - Paris
  - Pessac
  - Rennes
  - Strasbourg
  - Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Bourliere M, Bronowicki JP, de Ledinghen V, Hezode C, Zoulim F, Mathurin P, Tran A, Larrey DG, Ratziu V, Alric L, Hyland RH, Jiang D, Doehle B, Pang PS, Symonds WT, Subramanian GM, McHutchison JG, Marcellin P, Habersetzer F, Guyader D, Grange JD, Loustaud-Ratti V, Serfaty L, Metivier S, Leroy V, Abergel A, Pol S. Ledipasvir-sofosbuvir with or without ribavirin to treat patients with HCV genotype 1 infection and cirrhosis non-responsive to previous protease-inhibitor therapy: a randomised, double-blind, phase 2 trial (SIRIUS). Lancet Infect Dis. 2015 Apr;15(4):397-404. doi: 10.1016/S1473-3099(15)70050-2. Epub 2015 Mar 13. PMID 25773757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled study sites in France. The first participant was screened on 26 September 2013. The last study visit occurred on 12 November 2014.
Pre-assignment Details: 172 participants were screened.
Groups:
- LDV/SOF: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily plus placebo to match ribavirin (RBV) in a divided daily dose for 24 weeks
- LDV/SOF + RBV: Placebo to match LDV/SOF plus placebo to match RBV for 12 weeks, followed by LDV/SOF (90/400 mg) FDC tablet plus RBV (200 mg tablets) administered orally in a divided daily dose based on weight (1000 mg per day for participants weighing < 75 kg; 1200 mg per day for participants weighing ≥ 75 kg) for 12 weeks
Period: Overall Study
Arm/Group | LDV/SOF | LDV/SOF + RBV
Started | 78 | 77
Completed | 76 | 76
Not Completed | 2 | 1
Not completed — Lack of Efficacy | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- LDV/SOF: LDV/SOF (90/400 mg) FDC tablet once daily plus placebo to match RBV in a divided daily dose for 24 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF | LDV/SOF + RBV | Total
Number analyzed (Participants) | 78 | 77 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10.7) | 56 (7.4) | 56 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 56 | 58 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 76 | 75 | 151
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 1 | 4
  White | 75 | 76 | 151
Hepatitic C Virus (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.59) | 6.5 (0.47) | 6.5 (0.54)
HCV Genotype [Number; unit: participants]
  Genotype 1 (no confirmed subtype) | 1 | 1 | 2
  Genotype 1a | 50 | 48 | 98
  Genotype 1b | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, < 25 IU/mL) 12 weeks following the last dose of study drug.
  * 1 participant who was randomized to the LDV/SOF + RBV group who received placebo discontinued prior to receiving LDV/SOF + RBV and is excluded from the Full Analysis Set.
  * 1 participant who was randomized to the LDV/SOF + RBV group received LDV/SOF + placebo, and is counted in the LDV/SOF group for the safety analysis, and in the LDV/SOF+RBV group for the efficacy analysis (ie, in the Full Analysis Set).
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participant with genotype 1 HCV infection who were randomized and received at least 1 dose of active study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF | LDV/SOF + RBV
Number analyzed (Participants) | 77 | 77
percentage of participants | 97.4 | 96.1
Statistical Analysis 1: Comparison: LDV/SOF vs LDV/SOF + RBV; A sample size of 75 subjects in each treatment group would provide 80% power to detect a difference of 15% in SVR12 rates (80% vs 95%) between the 2 treatment groups; Test type: Superiority or Other; difference in proportions = 1.4, 95% CI 2-sided [-5.9 to 8.6] — The 2-sided 95% confidence interval (CI) on the difference in SVR12 rates between the 2 treatment groups was constructed based on stratum-adjusted Mantel-Haenszel (MH) proportions

2. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF | LDV/SOF + RBV
Number analyzed (Participants) | 77 | 77
percentage of participants
  SVR4 | 97.4 | 97.4
  SVR24 | 97.4 | 96.1

3. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ (ie, < 25 IU/mL) at Weeks 1, 2, 4, 8, 12, and 24
Time Frame: Weeks 1, 2, 4, 8, 12, and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF | LDV/SOF + RBV
Number analyzed (Participants) | 77 | 77
percentage of participants
  Week 1 | 7.8 | 9.1
  Week 2 | 50.6 | 59.7
  Week 4 | 97.4 | 97.4
  Week 8 | 98.7 | 100.0
  Week 12 | 100.0 | 100.0
  Week 24 | 100.0 | 100.0

4. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 8, and 12
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: Participants in Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF | LDV/SOF + RBV
Number analyzed (Participants) | 77 | 77
log10 IU/mL
  Week 1 (LDV/SOF: n = 75; LDV/SOF + RBV: n = 75) | -4.10 (0.558) | -4.27 (0.547)
  Week 2 (LDV/SOF: n = 77; LDV/SOF + RBV: n = 77) | -4.74 (0.926) | -4.94 (0.452)
  Week 4 (LDV/SOF: n = 77; LDV/SOF + RBV: n = 77) | -5.10 (0.582) | -5.19 (0.433)
  Week 8 (LDV/SOF: n = 77; LDV/SOF + RBV: n = 77) | -5.11 (0.597) | -5.20 (0.448)
  Week 12 (LDV/SOF: n = 77; LDV/SOF + RBV: n = 77) | -5.11 (0.595) | -5.20 (0.448)

5. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure is defined as
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Baseline to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF | LDV/SOF + RBV
Number analyzed (Participants) | 77 | 77
percentage of participants
  On-Treatment Virologic Failure | 0 | 0
  Virologic Relapse | 2.6 | 3.9

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Arm/Group | LDV/SOF | LDV/SOF + RBV
Serious Adverse Events (participants affected / at risk) | 8/78 | 4/77
Other Adverse Events (participants affected / at risk) | 67/78 | 72/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=78) | LDV/SOF + RBV (N=77)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Cranial nerve infection (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=78) | LDV/SOF + RBV (N=77)
Abdominal distension (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 5
Constipation (Gastrointestinal disorders) | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 8 | 14
Asthenia (General disorders) | 35 | 45
Fatigue (General disorders) | 15 | 7
Influenza like illness (General disorders) | 5 | 5
Bronchitis (Infections and infestations) | 13 | 4
Nasopharyngitis (Infections and infestations) | 5 | 4
Rhinitis (Infections and infestations) | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 8
Disturbance in attention (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 31 | 21
Insomnia (Psychiatric disorders) | 13 | 17
Irritability (Psychiatric disorders) | 9 | 7
Sleep disorder (Psychiatric disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 22
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Hypertension (Vascular disorders) | 7 | 7

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years